CLINICAL TRIAL: NCT03615755
Title: A Pilot Study of Short Duration Hyperbaric Oxygen Therapy to Improve HbA1c, Leukocyte, and Serum Creatinine in Patient With Diabetic Foot Ulcer Wagner 3-4
Brief Title: Short Duration Hyperbaric Oxygen Therapy to Improve HbA1c, Leukocyte, and Serum Creatinine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hendry Irawan (Other)
Responsible Party: Sponsor-Investigator, Hendry Irawan, Clinical Research, Udayana University
Organization: Udayana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HBOT_DFU
Record Dates: First submitted 2018-07-09; First posted 2018-08-06 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-05

CONDITIONS: Hyperbaric Oxygen Therapy; Diabetic Foot Ulcer; Type II Diabetes Mellitus
Keywords: Hyperbaric Oxygen Therapy; Diabetic Foot Ulcer; HbA1c; Leukocyte; Serum creatinine
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 2 | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Therapy (No Intervention): Standard Therapy (controlling blood sugar, antibiotic drug, ulcer debridement, wound care, offloading)
- Combination Therapy (Active Comparator): Standard Therapy with adjuvant Hyperbaric Oxygen Therapy (Total 10 sessions, each session used pressure 2.4 ATA for 90 minutes per day)
  Interventions: Other: Hyperbaric Oxygen Therapy (HBOT)

INTERVENTIONS:
Other: Hyperbaric Oxygen Therapy (HBOT) — The investigators used 10 sessions of HBOT. One session of HBOT uses oxygen at 2.4 ATA for 90 minutes per day at multiplace hyperbaric chamber. This therapy is given five sessions in a week, so it takes two weeks.
  Arms: Combination Therapy

SUMMARY:
The investigators want to evaluate the short duration HBOT can improve glycohemoglobin (HbA1c) levels, leukocyte count, and serum creatinine levels in patients with DFU (diabetic foot ulcer) Wagner 3-4.

DETAILED DESCRIPTION:
This study uses pretest and posttest control group design. All DM (diabetes mellitus) patients with DFU at Sanglah General Hospital, Denpasar who meet the inclusion and exclusion criteria and willing to follow the research procedure. All patients are signing the agreement paper after getting research explanation. All patients were briefed on the study research using HBOT. If the patients are willing to participate in the study and use HBOT was grouped to combination therapy, if the patients are willing to participate in the study but do not want to use HBOT was grouped to standard therapy, but if the patients are not willing participate then excluded.

All patients were taken blood test for HbA1c levels, leukocyte count, and serum creatinine levels before debridement, then grouped for standard therapy or standard therapy with 10 sessions of HBOT. One session of HBOT uses oxygen at 2.4 ATA (atmosphere absolute) for 90 minutes per day at multiplace hyperbaric chamber. This therapy is given five sessions in a week, so it takes two weeks. At the end of therapy, all blood tests were performed again in both groups.

The inclusion criteria were patients who had type 2 diabetes and DFU Wagner class 3 or 4, aged over 18 years, and underwent debridement with or without toe amputation. The exclusion criteria were patients who had severe organs dysfunction such as heart failure, pulmonary infection, pneumothorax, chronic obstructive pulmonary disease, and stroke.

Statistical analysis using SPSS 17.0 (SPSS Inc., Chicago, Illinois, USA). All variables were described before and after treatment. Analysis pretest and posttest values on both groups were used paired T-test and independent T-test. The statistical test results are significant if p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients who had type 2 diabetes and DFU Wagner class 3 or 4, aged over 18 years, and underwent debridement with or without toe amputation.

Exclusion Criteria:

* patients who had severe organs dysfunction such as heart failure, pulmonary infection, pneumothorax, chronic obstructive pulmonary disease, and stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
HbA1c levels | 2 weeks
  HbA1c levels test before the patients were done debridement (baseline) and after 2 weeks therapy.
Leukocyte count | 2 weeks
  Leukocyte count test before the patients were done debridement (baseline) and after 2 weeks therapy.
Serum creatinine | 2 weeks
  Serum creatinine levels test before the patients were done debridement (baseline) and after 2 weeks therapy.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kementerian Kesehatan Republik Indonesia. Diabetes Melitus Penyebab Kematian Nomor 6 di Dunia: Kemenkes Tawarkan Solusi Cerdik Melalui Posbind. (online) 2013 Sep. [cited 2016 Aug. 30] Available from: http://www.depkes.go.id/article/print/2383/diabetes-melitus-penyebab-kematian-nomor-6-di-dunia-kemenkes-tawarkan-solusi-cerdik-melalui-posbindu.html.
- [Background] Mendis S, Davis S, Norrving B. Organizational update: the world health organization global status report on noncommunicable diseases 2014; one more landmark step in the combat against stroke and vascular disease. Stroke. 2015 May;46(5):e121-2. doi: 10.1161/STROKEAHA.115.008097. Epub 2015 Apr 14. No abstract available. PMID 25873596
- [Background] Societe de Pathologie Infectieuse de Langue Francaise. Management of diabetic foot infections. Short text. Societe de Pathologie Infectieuse de Langue Francaise. Med Mal Infect. 2007 Jan;37(1):1-25. doi: 10.1016/j.medmal.2006.09.002. No abstract available. English, French. PMID 17357221
- [Background] World Health Organization. Global Report on Diabetes. Switzerland: WHO Press; 2016.
- [Background] Frykberg RG, Zgonis T, Armstrong DG, Driver VR, Giurini JM, Kravitz SR, Landsman AS, Lavery LA, Moore JC, Schuberth JM, Wukich DK, Andersen C, Vanore JV; American College of Foot and Ankle Surgeons. Diabetic foot disorders. A clinical practice guideline (2006 revision). J Foot Ankle Surg. 2006 Sep-Oct;45(5 Suppl):S1-66. doi: 10.1016/S1067-2516(07)60001-5. PMID 17280936
- [Background] Wounds International. International Best Practice Guidelines: Wound Management in Diabetic Foot Ulcers. London: Wounds International A division of Schofield Healthcare Media Limited Enterprise House; 2013.
- [Background] Kessler L, Bilbault P, Ortega F, Grasso C, Passemard R, Stephan D, Pinget M, Schneider F. Hyperbaric oxygenation accelerates the healing rate of nonischemic chronic diabetic foot ulcers: a prospective randomized study. Diabetes Care. 2003 Aug;26(8):2378-82. doi: 10.2337/diacare.26.8.2378. PMID 12882865
- [Background] Waniczek D, Kozowicz A, Muc-Wierzgon M, Kokot T, Swietochowska E, Nowakowska-Zajdel E. Adjunct methods of the standard diabetic foot ulceration therapy. Evid Based Complement Alternat Med. 2013;2013:243568. doi: 10.1155/2013/243568. Epub 2013 Jun 13. PMID 23843866
- [Background] Jeffcoate WJ, Game FL. Evidence for the use of biological therapies in ulcers of the foot in diabetes. BioDrugs. 2014 Feb;28(1):1-6. doi: 10.1007/s40259-013-0052-3. PMID 23832595
- [Background] Flood MS. Hyperbaric Oxygen Therapy for diabetic Foot Ulcers. The Journal of Lancaster General Hospital. 2007;2:140-145.
- [Background] Bhutani S, Vishwanath G. Hyperbaric oxygen and wound healing. Indian J Plast Surg. 2012 May;45(2):316-24. doi: 10.4103/0970-0358.101309. PMID 23162231
- [Background] Karadurmus N, Sahin M, Tasci C, Naharci I, Ozturk C, Ilbasmis S, Dulkadir Z, Sen A, Saglam K. Potential benefits of hyperbaric oxygen therapy on atherosclerosis and glycaemic control in patients with diabetic foot. Endokrynol Pol. 2010 May-Jun;61(3):275-9. PMID 20602302
- [Background] Aydin F, Kaya A, Karapinar L, Kumbaraci M, Imerci A, Karapinar H, Karakuzu C, Incesu M. IGF-1 Increases with Hyperbaric Oxygen Therapy and Promotes Wound Healing in Diabetic Foot Ulcers. J Diabetes Res. 2013;2013:567834. doi: 10.1155/2013/567834. Epub 2013 Feb 26. PMID 23671876
- [Background] El-Kader SMA, Ashmawy EM. Impact of Different Therapeutic Modalities on Healing of Diabetic Foot Ulcers. Eur J Gen Med. 2015;12:319-325.
- [Background] Gupta SK, Sharma AK. Effects of hyperbaric oxygen therapy on haematological and biochemical parameters. Ind J Aerospace Med. 2000;44:1-5.
- [Background] Al-Waili NS, Butler GJ, Beale J, Abdullah MS, Finkelstein M, Merrow M, Rivera R, Petrillo R, Carrey Z, Lee B, Allen M. Influences of hyperbaric oxygen on blood pressure, heart rate and blood glucose levels in patients with diabetes mellitus and hypertension. Arch Med Res. 2006 Nov;37(8):991-7. doi: 10.1016/j.arcmed.2006.05.009. PMID 17045116
- [Background] Nwafor TS, Collins N. Managing low blood glucose levels in patients undergoing hyperbaric oxygen therapy. Ostomy Wound Manage. 2014 Apr;60(4):12-5. No abstract available. PMID 24706399
- [Background] Wilkinson D, Chapman IM, Heilbronn LK. Hyperbaric oxygen therapy improves peripheral insulin sensitivity in humans. Diabet Med. 2012 Aug;29(8):986-9. doi: 10.1111/j.1464-5491.2012.03587.x. PMID 22269009
- [Background] Irawan H, Kartika. Terapi Oksigen Hiperbarik sebagai Terapi Adjuvan Kaki Diabetik. Cermin Dunia Kedokteran-245. 2016;43:782-785.
- [Background] Thom SR. Hyperbaric oxygen: its mechanisms and efficacy. Plast Reconstr Surg. 2011 Jan;127 Suppl 1(Suppl 1):131S-141S. doi: 10.1097/PRS.0b013e3181fbe2bf. PMID 21200283
- [Background] Klein KC, Guha SC. Cutaneous wound healing: Current concepts and advances in wound care. Indian J Plast Surg. 2014 Sep-Dec;47(3):303-17. doi: 10.4103/0970-0358.146574. PMID 25593414
- [Background] Mathieu D, Wattel F. Physiologic Effects of Hyperbaric Oxygen on Microorganisms and Host Defences Against Infection. In: Mathieu D, editor. Handbook on Hyperbaric Medicine. Netherlands: Springer; 2006. p.103-119.
- [Background] Wibowo A. Oksigen Hiperbarik: Terapi Percepatan Penyembuhan Luka. JuKe Unila. 2015;5:124-128.
- [Background] Uzun G, Mutluoglu M, Uz O. Hyperbaric oxygen therapy in diabetic patients - comments on the paper by Karadurmus et al. Endokrynol Pol. 2011;62(3):286-7. No abstract available. PMID 21717415
- [Background] Fife CE, Buyukcakir C, Otto G, Sheffield P, Love T, Warriner R 3rd. Factors influencing the outcome of lower-extremity diabetic ulcers treated with hyperbaric oxygen therapy. Wound Repair Regen. 2007 May-Jun;15(3):322-31. doi: 10.1111/j.1524-475X.2007.00234.x. PMID 17537119
- [Background] Kevin T. Pengaruh Terapi Oksigen Hiperbarik Terhadap eGFR berdasarkan Formula MDRD pada pasien Luka Kaki Diabetik (skripsi). Surabaya: Universitas Katolik Widya Mandala; 2015.
- [Background] Ayvaz S, Aksu B, Kanter M, Uzun H, Erboga M, Colak A, Basaran UN, Pul M. Preventive effects of hyperbaric oxygen treatment on glycerol-induced myoglobinuric acute renal failure in rats. J Mol Histol. 2012 Apr;43(2):161-70. doi: 10.1007/s10735-012-9391-5. Epub 2012 Feb 7. PMID 22311626
- [Background] Solmazgul E, Uzun G, Cermik H, Atasoyu EM, Aydinoz S, Yildiz S. Hyperbaric oxygen therapy attenuates renal ischemia/reperfusion injury in rats. Urol Int. 2007;78(1):82-5. doi: 10.1159/000096941. PMID 17192739
- [Background] Migita H, Yoshitake S, Tange Y, Choijookhuu N, Hishikawa Y. Hyperbaric Oxygen Therapy Suppresses Apoptosis and Promotes Renal Tubular Regeneration After Renal Ischemia/Reperfusion Injury in Rats. Nephrourol Mon. 2016 Jan 17;8(1):e34421. doi: 10.5812/numonthly.34421. eCollection 2016 Jan. PMID 26981502
- [Background] Rubinstein I, Abassi Z, Milman F, Ovcharenko E, Coleman R, Winaver J, Better OS. Hyperbaric oxygen treatment improves GFR in rats with ischaemia/reperfusion renal injury: a possible role for the antioxidant/oxidant balance in the ischaemic kidney. Nephrol Dial Transplant. 2009 Feb;24(2):428-36. doi: 10.1093/ndt/gfn511. Epub 2008 Sep 17. PMID 18799609
- [Background] Berkovitch M, Tsadik R, Kozer E, Abu-Kishk I. The effect of hyperbaric oxygen therapy on kidneys in a rat model. ScientificWorldJournal. 2014;2014:105069. doi: 10.1155/2014/105069. Epub 2014 Aug 10. PMID 25177712
- [Background] Singh VP, Bali A, Singh N, Jaggi AS. Advanced glycation end products and diabetic complications. Korean J Physiol Pharmacol. 2014 Feb;18(1):1-14. doi: 10.4196/kjpp.2014.18.1.1. Epub 2014 Feb 13. PMID 24634591
- [Derived] Irawan H, Semadi IN, Widiana IGR. A Pilot Study of Short-Duration Hyperbaric Oxygen Therapy to Improve HbA1c, Leukocyte, and Serum Creatinine in Patients with Diabetic Foot Ulcer Wagner 3-4. ScientificWorldJournal. 2018 Aug 12;2018:6425857. doi: 10.1155/2018/6425857. eCollection 2018. PMID 30158840

DOCUMENTS (3):
  • Study Protocol (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT03615755/Prot_003.pdf
  • Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT03615755/SAP_004.pdf
  • Informed Consent Form (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT03615755/ICF_005.pdf